CLINICAL TRIAL: NCT06686589
Title: The Utility of Hand-held Ultrasound Devices to Detect Bowel Wall Inflammatory Activity in Crohn's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Dr. Dan Carter, Gastroenterologist, Head, intestinal ultrasound service, Sheba Medical Center
Other Study IDs: SHEBA-23-0523-DC-CTIL
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Crohn Disease (CD)
Keywords: Crohn disease; intestinal ultrasound; hand held ultrasound
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn's patients undergoing routine intestinal ultrasound exam
  Interventions: Diagnostic Test: Intestinal ultrasound

INTERVENTIONS:
Diagnostic Test: Intestinal ultrasound — Intestinal ultrasound performed by hand held ultrasound devices

SUMMARY:
One of the major obstacles in implementing intestinal ultrasound services for inflammatory bowel disease (IBD) patients relates to the costs of acquiring ultrasound (US) machines. The costs of high-end (and higher levels of quality) US machines are considerable, and although large medical centers in developed countries can obtain US machines, smaller centers in rural areas, community centers and centers in undeveloped countries may struggle with the cost of the machines. The lack of availability of point-of-care intestinal ultrasound impedes the medical treatment IBD patients receive. Recently, new models of hand-held small ultrasound machines were introduced to the market by large ultrasound companies. These machines are affordable and are used mainly for point-of-care ultrasound exams. We hypothesize that if the image quality acquired by these machines is proven to be good enough for the detection of bowel inflammation and complications in Crohn's disease (CD) patients, the use of intestinal ultrasound can potentially increase, allowing better care for CD patients.

Our idea is to compare the accuracy of various hand-held ultrasound devices to detect ultrasonographic signs of bowel inflammatory activity (especially increased bowel wall thickness) to that of high-end and premium US machines. The first part of the project will include examining the quality of 2 different hand-held US machines (GE VSCAN air and Philips Lumify) by 3 experienced ultra-sonographers. If the achieved level of accuracy for the detection of bowel wall inflammatory activity will be sufficient (AUC>0.8), we aim to move to the second part of the project. This step focuses on hand-held US machines by gastroenterologists with various levels of IUS experience. Therefore, we aim to examine the accuracy of hand-held US machines for the detection of inflammatory activity by delivering the hand-held US machines to 10 GI specialists who completed the IBUS educational curriculum for IUS (at least module 1+2) with various levels of IUS expertise.

* Project Goal 1) To examine the capability and accuracy of hand-held ultrasound machines to detect bowel wall inflammatory activity and complications in CD patients.
* Strategy - Comparing various ultrasonographic signs of inflammation acquired by hand-held US machines to that acquired by high-end and premium US machines.
* Outcomes - Accuracy of hand-held ultrasound machines in the detection of bowel wall inflammatory activity The problem being addressed by the proposed project - Dissemination of IUS is limited due to the high costs of US machines. The use of affordable hand-held US machines for the detection of inflammatory activity will expand the IUS incorporation into the CD diagnosis, monitoring, and treatment approaches, improving patient outcomes.

Significance/Impact The use of affordable and precise US machines will disseminate the use of IUS and expand the IUS incorporation into the diagnosis, monitoring, and treatment of CD, improving patient outcomes

DETAILED DESCRIPTION:
• Aim 1. Comparison of the accuracy of hand-held US machines for the detection and measurement of bowel wall inflammatory activity to that of advanced high-end and premium US machines by experienced IUS performers

* Rationale: IUS use has been incorporated into the processes of diagnosis, follow-up, monitoring, and treatment approaches in CD. One of the limiting factors of IUS dissemination relates to the high costs of the modern high-end and premium US machines used for intestinal ultrasound. Confirming the acceptable accuracy of affordable modern hand-held US machines for detection and measurement of inflammatory activity will enable dissemination of IUS use, as obtaining affordable and precise US machines will be possible.
* Overall Experimental Strategy and/or Methodology: 150 CD patients will undergo an IUS exam using a hand-held US machine (GE VSCAN air or Philips Lumify) followed by an exam using a high-end or premium US machine (GE S-8, BK 3000 and GE E-9). All exams will be performed by one of 3 experienced IUS performers (DC, AA, HB). The exams will be performed using the same consecutive method with a low-frequency curved array transducer enabling all abdominal quadrants to be examined for fill levels, potential pathological distension, motility, and para-intestinal structures such as abscesses, followed by examination using a high-resolution linear array for detailed examination of the bowel wall structure. All examinations will be performed without any preceding preparation, using a consistent technique and protocol, beginning the examination with the terminal ileum (TI), proximal to the distal colon, followed by an examination of the small bowel. The assessment will be performed for features of inflammation, especially bowel wall thickness of the TI and the colon. Bowel wall thickness will be measured at least in two different areas at a minimal distance of 1 cm from each other. Colonic bowel thickness will be measured at the right, transverse, left, and sigmoid colon. Small bowel wall thickness will be measured at the TI. The thickest measurement of each bowel segment will be chosen as a representative for measurement. Images and cine-loops of each segment of the colon and the TI will be saved on the tablet connected to the hand-held US machine.

Other signs of inflammation will also be examined: Doppler signs within the bowel wall using the modified Limberg scoring system, mesenteric fat hypertrophy, stratification of bowel wall layers and enlargement of lymph nodes.

Intramural and extramural complications including strictures with\without pre-stenotic dilatations, fistulas, and abscesses will be noted and the relative images will be saved.

The findings of different signs of inflammation described will be compared between the hand-held ultrasound and the high-end \ premium US machines. A dichotomic comparison for the presence of each sign (yes/no) will be followed by a comparison of numerical parameters (exact bowel thickness measurement for each segment and Limberg score).

* The saved images and cine loops of each segment will be reviewed blindly by one of the other sonographers and assessed for inter-reader agreement between different performers.
* An ICC analysis will be performed for the primary outcome of bowel wall thickness.
* Expected Outcomes/Results: To define if the hand-held US machine can detect basic ultrasonographic signs of inflammation (bowel wall thickness) with adequate accuracy compared with gold-standard high-end \ premium US machines.

  • Aim 2: Comparison of the accuracy of hand-held US machines for the detection and measurement of bowel wall inflammatory activity to that of advanced high-end and premium US machines by ultra-sonographers with ultra-sonographers with various experience levels.
* Rationale: Judging from preliminary experience, we hypothesize hand-held US machines will be accurate for the detection of inflammatory activity when used by experienced IUS performers. However, the accuracy of the hand-held ultrasound machine used by less experienced users will still need to be verified.
* Overall Experimental Strategy and/or Methodology:

Different levels of IUS experience will be defined based on the time from the conclusion of the IBUS curriculum and the number of IUS exams performed per month:

Novice- up to one year after the conclusion of the IBUS curriculum. Performs at least 20 exams per month.

Intermediate experience- 1-2 years after the conclusion of the IBUS curriculum. Performs at least 20 exams per month. Total exams performed 500-1000 Experienced- >2 years after the conclusion of the IBUS curriculum. Performed> 1000 exams.

* Hand-held ultrasound machines will be used by 10 ultra-sonographers with different levels of experience (3 novices, 4 intermediates, 3 experienced). The first 20 exams will be performed for reaching confidence using the US machine. Each ultra-sonographer will perform 50 exams using hand-held US machines and compare the results to the following exam performed by a high-end \ premium US machine (the same machines used for IUS in every sonographer's hospital). The assessment will be performed for features of inflammation, especially bowel wall thickness of the TI and the colon. Bowel wall thickness will be measured at least in two different areas at a minimal distance of 1 cm from each other. Colonic bowel thickness will be measured at the right colon, transverse colon, left colon and sigmoid colon. Small bowel thickness will be measured at the TI. The thickest segment of each bowel segment will be chosen for the purpose of measurement. Images and cine-loops of each segment of the colon and the TI will be saved on the tablet connected to the hand-held US machine. Other signs of inflammation will also be examined: Doppler signs within the bowel wall using the modified Limberg scoring system, fat hypertrophy, stratification of bowel wall layers and enlargement of lymph nodes. Intramural and extramural complications including strictures with\without pre-stenotic dilatations, fistulas and abscesses will be noted and the relative images will be saved. The findings of different signs of inflammation described will be compared between the hand-held ultrasound and the high-end \ premium US machines. Dichotomic comparison for the presence of each sign (yes/no) will be followed by a comparison of numerical parameters when possible (exact bowel thickness measurement for each bowel segment and Limberg score). Intramural and extramural complications including strictures with\without pre-stenotic dilatations, fistulas and abscesses will be noted and the relative images will be saved. The findings of different signs of inflammation described will be compared between the hand-held ultrasound and the high-end \ premium US machines.
* 20 percent of each performer's saved images and cine loops will be reviewed blindly by one of the 3 expert sonographers and assessed for the inter-reader agreement between performers.

ELIGIBILITY:
Inclusion Criteria:

Crohn disease of the terminal ileum and colon- Age> 18

Exclusion Criteria:

* Pregnancy Inability to visualize he bowel on US Proximal Crohn's disease Proctitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 150 consecutive Crohn's patients going through intestinal ultrasound at the discretion of their referring physician.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The capability and accuracy of hand-held ultrasound machines to detect bowel wall inflammatory activity and complications in CD patients. | fro enrollmeent to the end of the study at 2 years
  Comparing various ultrasonographic signs of inflammation acquired by hand-held US machines to that acquired by high-end and premium US machines. Defining accuracy of hand-held ultrasound machines in the detection of bowel wall inflammatory activity

CONTACTS AND LOCATIONS:
Overall Officials: Dan Carter, Associate Professor, Principal Investigator — Sheba Medical Center

IPD SHARING:
Plan to Share IPD: No
IUS images - the data for he study- can not be shared due to patient privecy issure

DOCUMENTS (1):
  • Study Protocol (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT06686589/Prot_000.pdf